CLINICAL TRIAL: NCT00362583
Title: A Double-blind, Randomised, Placebo-controlled Trial Confirming the Efficacy of Intranasal Fentanyl Titrated to 50, 100 or 200 µg With an Open Long-term Safety Follow-up in Cancer Patients With Breakthrough Pain
Brief Title: Efficacy and Safety of Intranasal Fentanyl in the Treatment of Breakthrough Pain (FT-018-IM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FT-018-IM; 2005-002348-24
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Cancer
Keywords: Cancer pain with breakthrough pain episodes
MeSH Terms: conditions — Neoplasms | interventions — Fentanyl

INTERVENTIONS:
Drug: Fentanyl

SUMMARY:
Primary objectives:

* To confirm the efficacy of intranasal fentanyl titrated to doses 50, 100 or 200 µg for treatment of breakthrough pain (BTP) in cancer patients
* To establish long-term safety of treatment with intranasal fentanyl

Secondary objectives:

- To explore the relationship between dose of background opioid treatment and titrated fentanyl dose

ELIGIBILITY:
Inclusion Criteria:

1. Has the patient given informed consent according to local requirements before any trial-related activities? Trial-related activities are any procedure that would not have been performed during the routine management of the patient
2. Is the patient a cancer patient with breakthrough pain?
3. Is the patient aged ≥18 years?
4. Has the patient received for at least the past month either oral morphine, oxycodone, hydromorphone or transdermal fentanyl for treatment of background pain?
5. Is the current dose of the scheduled background opioid of the patient equivalent to 60-500 mg oral morphine/day or to transdermal fentanyl 25-200 µg/hour? For conversion table.
6. Is the background pain generally stable and on average controlled to a mild level (defined as ≤4 on an 11 point NRS) by the background opioid?
7. Is the BTP(s) in general of so severe pain intensity that the patient judges he/she needs additional analgesics (apart from background pain analgesics) and does it normally last for more than 15 minutes?
8. Does the patient in general while using a stable, fixed-schedule, opioid regimen have at least three BTP episodes per week but no more than four BTP episodes per day?*
9. Has the patient obtained at least partial relief of BTP(s) with his/her usual immediate-release strong opioid, i.e. oral morphine, oxycodone, hydromorphone or transmucosal fentanyl?
10. Is the patient able to use intranasal drugs?
11. Does the patient use adequate contraceptive precaution (contraceptive pill, implant or injection or intrauterine device) in the trial period?
12. Did the patient have a negative pregnancy test at the inclusion in studies FT-016-IM or FT-017-IM?

Exclusion Criteria:

All exclusion criteria must be answered "no" for a patient to participate in the trial.

1. Does the patient have a recent history of substance abuse?
2. Is the patient pregnant or nursing during the trial period?
3. Has the patient neurological or psychiatric impairment that may compromise data collection?
4. Has the patient severe hepatic impairment? (Investigator's judgement according to local practice)
5. Has the patient had any recent therapy, which could potentially alter pain or response to analgesics to a degree, where the need for background opioid will be less than 60 mg morphine or morphine equivalents/day or less than 25 µg/hour transdermal fentanyl or the number of BTP episodes will be less than three per week during the trial period?
6. Has the patient had facial radiotherapy?
7. Has the patient been treated with MAO inhibitor within the last 14 days?
8. Does the patient use Methadone or Buprenorphine?
9. Does the patient have an impaired respiratory function to an extent, which may severely increase the risk of clinically relevant respiratory depression by BTP fentanyl treatment?
10. Does the patient use drugs for intranasal administration?
11. Does the patient have nasopharyngeal probe?
12. Is the patient known to be hypersensitive to fentanyl or to other opioids or any of their excipients?
13. Has the patient any head injury, primary brain tumour or other pathological conditions, which could significantly increase the risk of increased intracranial pressure or impaired consciousness?
14. Has the patient concomitant participation in any other trial with an investigational drug or device apart from cancer treatment and participation in intranasal fentanyl trials FT-016-IM/ FT-017-IM within 30 days prior to inclusion in this trial?
15. Does the patient have pathological conditions of the nasal cavity as contraindication to intranasal fentanyl?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark